CLINICAL TRIAL: NCT06560645
Title: A Phase 1 Open-Label, Multi-Center, Safety and Efficacy Study of PRT7732, an Oral SMARCA2 Degrader, in Patients With Advanced or Metastatic Solid Tumors With a SMARCA4
Brief Title: A Study of PRT7732, an Oral SMARCA2 Degrader, in Patients With Advanced or Metastatic Solid Tumors With a SMARCA4 Mutation
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Prelude Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRT7732-01
Record Dates: First submitted 2024-08-06; First posted 2024-08-19 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumor; Metastatic Solid Tumor; Non-small Cell Lung Carcinoma; SMARCA4 Mutation; Esophageal Adenocarcinoma; Esophageal Squamous Cell Carcinoma; Gastric Adenocarcinoma; Gastric Squamous Cell Carcinoma; Gastroesophageal Junction Adenocarcinoma; Gastroesophageal Junction Squamous Cell Carcinoma
Keywords: Advanced Solid Tumors; BRG1; BRM; Degrader; Metastatic Solid Tumors; Non-Small Cell Lung Cancers; NSCLC; PRT7732; SMARCA2; SMARCA4; Esophageal Adenocarcinoma; Esophageal Squamous Cell Carcinoma; Gastric Adenocarcinoma; Gastric Squamous Cell Carcinoma; Gastroesophageal Junction Adenocarcinoma; Gastroesophageal Junction Squamous Cell Carcinoma
MeSH Terms: conditions — Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PRT7732 (Experimental): PRT7732 is administered as an oral capsule once daily. Dose escalation/de-escalation decisions will be guided by the BLRM method until the RDE is determined.
  Interventions: Drug: PRT7732

INTERVENTIONS:
Drug: PRT7732 — PRT7732 capsules will be self-administered once daily at the dose-level assigned

SUMMARY:
This is a Phase 1 study to determine the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary efficacy of PRT7732 in patients with select advanced or metastatic solid tumors with a SMARCA4 mutation.

DETAILED DESCRIPTION:
This is an open-label, multi-center, first-in-human, Phase 1 study to determine the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary efficacy of PRT7732 an oral SMARCA degrader in patients with select advanced or metastatic solid tumors with a SMARCA4 mutation. Approximately 104 participants will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations (including contraception requirements), and other study procedures
* Histologically confirmed advanced, recurrent, or metastatic solid tumor malignancy with any mutation of SMARCA4 by local testing that has either progressed on or is ineligible for standard of care therapy
* Must have measurable or non-measurable (but evaluable) disease per RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Willing to provide either archival or fresh tumor tissue sample
* Adequate organ function (hematology, renal, and hepatic)

Exclusion Criteria:

* Participants with solid tumors with known concomitant SMARCA2 mutation or loss of protein expression
* Clinically significant or uncontrolled cardiac disease, uncontrolled electrolyte disorders, uncontrolled or symptomatic central nervous system (CNS) metastases or leptomeningeal disease
* History of other malignancy within 3 years except for adequately treated basal cell or squamous cell skin cancer, superficial bladder cancer, prostate intraepithelial neoplasm, prostate adenocarcinoma with Gleason score of 3+3 or less, carcinoma in situ of the cervix, or other non-invasive or indolent malignancies, or malignancies previously treated with curative intent and not on active therapy or expected to require treatment or recurrence during the study
* Receipt of any targeted therapy directed against BRM/BRG1 (SMARCA2/SMARCA4).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-11-04 (Actual); Primary Completion 2026-01-28 (Actual); Study Completion 2026-01-28 (Actual)

PRIMARY OUTCOMES:
Dose Limiting toxicity (DLT) of PRT7732 | Baseline through Day 21
  Incidence of dose limiting toxicities for patients in the dose escalation phase
Safety and tolerability of PRT7732 as measured by incidence of DLTs | Baseline through completion of study, an average of 2 years
  Safety and tolerability will be evaluated by incidence of DLTs
Safety and tolerability of PRT7732 as measured by incidence of laboratory deviations | Baseline through study completion, an average of 2 years
  Safety and tolerability will be evaluated by laboratory measurements
Safety and tolerability as measured by rates of dose modification due to AEs according to NCI CTCAE | Baseline through study completion, an average of 2 years
  Safety and tolerability will be evaluated by dose interruption, modification, and discontinuation due to adverse events (AEs) according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE)
Maximum tolerated dose (MTD) of PRT7732 | Baseline through study completion, an average of 2 years
  Maximum tolerated dose will be determined by the sponsor based on the Safety Review Committee's recommendation considering the totality of the available clinical safety, clinical efficacy, pharmacokinetics (PK), and pharmacodynamic data
Recommended dose for expansion (RDE) of PRT7732 | Baseline through study completion, an average of 2 years
  The RDE will be determined by the sponsor based on the Safety Review Committee's recommendation considering the totality of the available clinical safety, clinical efficacy, pharmacokinetics (PK), and pharmacodynamic data

SECONDARY OUTCOMES:
Efficacy of PRT7732 | Baseline through study completion, an average of 2 years
  Best overall response of either complete response (CR) or partial response (PR), as assessed by the investigator per RECIST v1.1
Pharmacokinetic profile of PRT7732 as a single agent: Maximum observed plasma concentration | Baseline through study completion, an average of 2 years
  Pharmacokinetics will be calculated including the maximum observed plasma concentration
Pharmacokinetic profile of PRT7732 as a single agent: Area under the curve | Baseline through study completion, an average of 2 years
  Pharmacokinetics will be calculated including the area under the plasma concentration versus time curve (AUC)
Pharmacokinetic profile of PRT7732 as a single agent: Time of maximum concentration (Tmax) and half-life (T1/2) | Baseline through study completion, an average of 2 years
  Pharmacokinetic parameters will be calculated using standard non-compartmental techniques
Pharmacodynamic effects of PRT7732 as a single agent | Baseline through study completion, an average of 2 years
  The pharmacodynamic effect of PRT7732 demonstrating target engagement by assessment of SMARCA2 protein in peripheral blood mononuclear cells and tumor tissue as assessed by reduction in protein levels of SMARCA2 in peripheral blood mononuclear cells and/or tumor tissue

CONTACTS AND LOCATIONS:
Locations (28):
- United States (11):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Brigitte Harris Cancer Pavilion, Detroit, Michigan
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Memorial Sloan Kettering Cancer Center - Main Campus, New York, New York
  - UNC Hospitals, The University of North Carolina Chapel Hill, Chapel Hill, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - SCRI Oncology Partners, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Virginia Comprehensive Cancer Center, Charlottesville, Virginia
- Australia (5):
  - Border Medical Oncology Research Unit, Albury, New South Wales
  - Southern Highlands Cancer Centre, Bowral, New South Wales
  - Scientia Clinical Research Ltd, Randwick, New South Wales
  - Monash Health, Clayton, Victoria
  - Linear Clinical Research Ltd, Nedlands, Western Australia
- Germany (2):
  - University Clinic Cologne, Clinic for Internal Medicine, Cologne, North Rhine-Westfalia
  - Technische Universitat Dresden, Medizinlsche Fakultat Carl Gustav Carus Nationales Centrum fur Tumorerkrankungen Dresden, Early Clinical Trial Unit (NCT/UCC ECTU), Dresden, Saxony
- Japan (4):
  - Kindai University Hospital, Sayama, Osaka
  - The Univerity of Osaka Hospital, Suita, Osaka
  - National Cancer Center Hospital, Chuo Ku, Tokyo
  - Cancer Institute Hospital of JFCR, Koto-ku, Tokyo
- South Korea (3):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
- Spain (3):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Start Madrid-FJD, Hospital Universitario Fundacion Jimenez Diaz-Servicio de Oncologia, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid